CLINICAL TRIAL: NCT06018272
Title: Mentalisierungsbasierte Therapie Versus Bona-fide-Therapie für Patient:Innen Mit Borderline-Persönlichkeitsstörung in Deutschland (MaGnet): Eine Prospektive, Multizentrische Randomisiert-kontrollierte Studie Mentalization-based Treatment Versus Bona-fide Treatment for Patients With Borderline Personality Disorder in Germany (MAGNET): a Prospective, Multi-centre Randomized Controlled Trial
Brief Title: Mentalization-based Treatment Versus Bona-fide Treatment for Patients With Borderline Personality Disorder in Germany
Acronym: MAGNET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Research Foundation (Other); University Düsseldorf (Other); Jena University Hospital (Other); Universitätsklinikum Ulm (Unknown); Psychologische Hochschule Berlin (Unknown)
Responsible Party: Principal Investigator, Svenja Taubner, Prof. Dr. phil. Svenja Taubner, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 500412881
Record Dates: First submitted 2023-08-17; First posted 2023-08-30 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentalization-Based Treatment (MBT) (Experimental)
  Interventions: Behavioral: Mentalization-Based Treatment (MBT)
- Bona-Fide Treatment in Germany (BFT) (Active Comparator)
  Interventions: Behavioral: Bona-Fide Treatment in Germany (BFT)

INTERVENTIONS:
Behavioral: Mentalization-Based Treatment (MBT) — Patients in MBT will receive a maximum of 58 sessions in total. Of those, 30 are weekly individual sessions. 28 sessions are weekly group sessions conducted by two therapists, and consisting of 8 introductory sessions of group psychoeducation followed by 20 group therapy sessions. The duration of MBT is 12 months. MBT is manualized and relies on validating the emotional experience of patients that aims to promote mentalizing. The proposed mechanism of change in MBT is to stabilize mentalizing in certain focus areas in order to create a psychic buffer between affect and behaviour to foster affect regulation, reduce impulsivity and promote functional supportive relationships.
  Arms: Mentalization-Based Treatment (MBT)
Behavioral: Bona-Fide Treatment in Germany (BFT) — Patients in BFT will receive one to two weekly sessions of Bona-Fide-Treatment (Psychodynamic Therapy, PT, or Cognitive Behavioural Therapy, CBT) conducted by community experts delivered as short-term psychotherapy (<24 sessions) or long-term psychotherapy (>24 sessions). BFT can be delivered as individual, group or a combination of individual and group treatment as stated in the German psychotherapy regulations.
  Arms: Bona-Fide Treatment in Germany (BFT)

SUMMARY:
Background: Borderline Personality Disorder (BPD) is a serious mental disorder. Mentalization-based treatment (MBT) is one evidence-based treatment for individuals with BPD. Specifically, MBT has been highlighted for its effectiveness in reduction of suicidal and non-suicidal self-injury (NSSI). Yet, randomized-controlled trials (RCT) on MBT in outpatient settings compared with bona fide treatment (BFT) are still scarce and none has been conducted in Germany. The primary objective of this RCT is to investigate whether outpatient MBT is more effective in the reduction of crisis events (incidences of NSSI and suicide attempts) compared with BFT (namely psychodynamic or cognitive-behavioural psychotherapy) in Germany. Secondary, MBT's efficacy will be investigated with regard to cost-effectiveness, general and interpersonal functioning, BPD and general symptom severity, social adjustment, quality of life, reduction in psychotropic medication and therapy retention. Additionally, moderator as well as common and treatment specific mediator variables will be investigated.

Study Design/ Study Population/ Methods: Across 5 study sites in Germany, 304 individuals of all genders from age 18 to 65 with a BPD diagnosis and NSSI or suicide attempts in the past will be asked to participate in the study for two years. In the first year, patients will receive either MBT or BFT (psychodynamic or cognitive behavioural psychotherapy) and will take part in continuous scientific assessments. Scientific assessments will continue after therapy completion up to a 12-moth follow up. As primary outcome, crisis events will be assessed via ecological momentary assessment (EMA) four times a week once per month during the first year and once every three months in the second year. Number of crisis events up to 2 years post randomization will be compared between treatment arms using a log-linear regression model following an intention-to-treat approach. Secondary outcomes, such as borderline and general symptom severity, will be assessed at several timepoints. A within-trial cost-effectiveness analysis (CEA) will be conducted with a societal perspective.

Clinical Trial Rationale: This study investigates efficacy of MBT as BPD specific treatment in an outpatient setting compared with BFT in Germany. Results of this study can address a treatment gap in the German healthcare system, and inform about health economic aspects of BPD treatment as well as mechanisms of psychotherapeutic change.

ELIGIBILITY:
Inclusion Criteria:

* Borderline Personality Disorder
* non-suicidal self injury or suicide attempts in the past two years as indicated by the IPDE item "repeated suicidal behaviours, gestures, threats or self-harm", one of which has occurred in the past six months

Exclusion Criteria:

* acute substance use disorder (exception: cannabis dependency)
* diagnosis of schizophrenia or schizotypal personality disorder
* bipolar I disorder (DSM-5)
* cognitive impairment (IQ<80) or evidence of organic brain disorder
* BMI<16.5
* serious medical condition that will require hospitalization within the next year (e.g. cancer)
* no sufficient German language abilities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
change in crisis events assessed with Ecological Momentary Assessment with items based on the SHBQ (Gutierrez et al., 2001) | every second day during one week per month in the first year, and during one week every three months in the second year
  composite score (non)suicidal self injury

SECONDARY OUTCOMES:
Symptoms of Borderline Personality Disorder assessed with the IPDE (Loranger et al., 1997) and BSL-23 (Wolf et al., 2009) | Day 0, Month 6, Month 12, Month 24; IPDE only at Month 24
Change in psychiatric symptom severity assessed with the DASS- 21 (Lovibond & Lovibond, 1995) | Day 0, Month 6, Month 12, Month 24
Change in health and disability assessed with WHODAS 2.0 Short Form (Üstün et al., 2010) | Day 0, Month 6, Month 12, Month 24
Change in personality funcitioning assessed with LPFS-BF (Hutsebaut et al., 2016) | Day 0, Month 6, Month 12, Month 24
Change in personality traits assessed with PID5BF+M (Bach et al., 2020) | Day 0, Month 6, Month 12, Month 24
Change in threat hypersensitivity assessed with emotion classification task (Honecker et al., 2021) | Day 0, Month 6, Month 12, Month 24
  Participants are presented with 160 faces, each unambiguously showing one of four emotional expressions (angry, fearful, happy, neutral). The goal of the task is to correctly classify these facial expressions. The task's collected behavioral data encompasses two key measurements: the ratio of accurate responses (specifically, correct emotion classification) and the time it takes to respond in trials where the emotion classification is correct.
Change in quality of life assessed with EQ-5D-5L (Herdman et al., 2011; EuroQol Research Foundation, 2019) | Day 0, Month 6, Month 12, Month 24
Change in trait anger assessed with STAXI-2 (Spielberger, 1999) | Day 0, Month 6, Month 12, Month 24
Change in social adjustment assessed with WSAS (Marks, 1986) | Day 0, Month 6, Month 12, Month 24
Change in emotional reactions to social exclusion, rejection and relational devaluation with SPQ (Stangier et al., 2021) | Day 0, Month 6, Month 12, Month 24
Change in Interoceptive Body Awareness with MAIA-2 (Mehling et al., 2018) | Day 0, Month 6, Month 12, Month 24
Changes in medication with self-report of medication prescription via adapted version of AD-SUS (Kuyken et al., 2015) | Day 0, Month 6, Month 12, Month 24
Heath Care utilization with an adapted version of the AD-SUS (Kuyken et al., 2015) | Day 0, Month 6, Month 12, Month 24
Change in acute dissociative symptoms with Dissociation-Tension Scale-4 (DSS-4; Stiglmayr et al., 2003) | Day 0, Month 6, Month 12, Month 24

OTHER OUTCOMES:
Mentalizing as mediator of change assessed with the Certainty About Mental States Questionnaire (CAMSQ; Müller et al., 2021) | Month 6, Month 12
  Mediator
Therapeutic Agency Inventory (TAI; Huber et al., 2019) | once a week in the first year and at Month 6 and Month 12
  Mediator
Group Questionnaire - short (GQ; Jensen, 2016) | once a week in the first year and at Month 6 and Month 12
  Mediator
Epistemic Trust, Mistrust and Credulity Questionnaire (ETMCQ; Campbell et al., 2019) | Month 6, Month 12
  Mediator
Experiences in Close Relationships-Revised Screening Version (ECR-RD8; Ehrenthal et al., 2021) | Month 6, Month 12
  Mediator
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Month 6, Month 12
  Mediator
Mentalizing as mediator of change assessed with Mentalizing Emotions Questionnaire (Kasper et al., submitted) | Month 6, Month 12
  Mediator
Negative Effects Questionnaire (NEQ; Rozental et al., 2016) | Month 12
  Serious adverse events of therapy
Therapeutic Alliance as mediator of change assessed with Working Alliance Inventory (WAI-SR, Hatcher & Gillaspy, 2006) | once a week in the first year and at Month 6 and Month 12
  Mediator
Symptoms of PTSD and complex PTSD and complex PTSD Trauma experiences with Internation Trauma Interview (ITI; Roberts et al., 2019) | Day 0
  Moderator
Symptoms of PTSD and complex PTSD with International Trauma Questionnaire (ITQ; Cloitre et al., 2018) | Day 0
  Moderator
Level of personality functioning with Semi-Structured Interview for Personality Functioning DSM-5 (STiP; Hutsebaut et al., 2017) | Day 0
  Moderator
Change of pleasure, arousal and dominance with Self-Assessment Manikin (Bradley, 1994) | once a week in the first year and at Month 6 and Month 12
  Mediator
Change of frequency of occurence of positive and negative automatic thoughts with Automatic Thoughts Questionnaire - Revised (ATQ-R; Kendall, 1989) | Month 6, Month 12
  Mediator
Assessment of the frequency of alliance ruptures and resolution processes in therapy sessions with Rupture Resolution Rating System (Eubanks et al., 2015) | Month 6, Month 12
  Mediator
Assessment of the clients'attachment style with the Patient Attachment Coding System (Talia & Miller-Bottome, 2012) | Month 6, Month 12
  Mediator
Assessment of the therapists' attunement and attachment status with the Therapist Attunement Scales (Talia & Muzi, 2017) | Month 6, Month 12
  Mediator
Assessment of the therapists' activity and appropriateness in essential domains of MBT with the Mentalization-Based Treatment Adherence and Competence Scale (Bateman & Fonagy, 2016) | Month 6, Month 12
  Mediator
Assessment of the therapists' adherence to psychodynamic-interpersonal and cognitive-behavioural treatments with the Comparative Psychotherapy Process Scale (Hilsenroth et al., 2005) | Month 6, Month 12
  Mediator
Interview for treatment and study evaluation | Month 24
  Semi-structured interview developed based on Krause et al. 2016 will be used to assess how patients experienced the therapy and the study, what aspects they perceived as positive or negative, and what impact the therapy had on their symptoms and their life

CONTACTS AND LOCATIONS:
Overall Officials: Svenja Taubner, Principal Investigator — University Heidelberg
Locations (5):
- Germany (5):
  - Psychologische Hochschule Berlin, Berlin
  - Clinic for Psychosomatic Medicine and Psychotherapy, University Hospital Düsseldorf, Düsseldorf
  - Heidelberg University, Heidelberg
  - Institute for Psychosocial Medicine, Psychotherapy and Psychooncology, Jena
  - Clinic for Psychosomatic Medicine and Psychotherapy, University Hospital Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bateman A, Fonagy P. Mentalization based treatment for borderline personality disorder. World Psychiatry. 2010 Feb;9(1):11-5. doi: 10.1002/j.2051-5545.2010.tb00255.x. PMID 20148147
- [Background] Bateman A, Fonagy P. Effectiveness of partial hospitalization in the treatment of borderline personality disorder: a randomized controlled trial. Am J Psychiatry. 1999 Oct;156(10):1563-9. doi: 10.1176/ajp.156.10.1563. PMID 10518167
- [Background] Bateman A, Fonagy P. Randomized controlled trial of outpatient mentalization-based treatment versus structured clinical management for borderline personality disorder. Am J Psychiatry. 2009 Dec;166(12):1355-64. doi: 10.1176/appi.ajp.2009.09040539. Epub 2009 Oct 15. PMID 19833787
- [Background] Jorgensen CR, Freund C, Boye R, Jordet H, Andersen D, Kjolbye M. Outcome of mentalization-based and supportive psychotherapy in patients with borderline personality disorder: a randomized trial. Acta Psychiatr Scand. 2013 Apr;127(4):305-17. doi: 10.1111/j.1600-0447.2012.01923.x. Epub 2012 Aug 17. PMID 22897123
- [Background] Laurenssen EMP, Luyten P, Kikkert MJ, Westra D, Peen J, Soons MBJ, van Dam AM, van Broekhuyzen AJ, Blankers M, Busschbach JJV, Dekker JJM. Day hospital mentalization-based treatment v. specialist treatment as usual in patients with borderline personality disorder: randomized controlled trial. Psychol Med. 2018 Nov;48(15):2522-2529. doi: 10.1017/S0033291718000132. Epub 2018 Feb 26. PMID 29478425
- [Background] Rossouw TI, Fonagy P. Mentalization-based treatment for self-harm in adolescents: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2012 Dec;51(12):1304-1313.e3. doi: 10.1016/j.jaac.2012.09.018. PMID 23200287
- [Background] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Result] Wittchen H-U, Zaudig M, Fydrich T. Strukturiertes Klinisches Interview für DSM-IV (SKID I und SKID II). Göttingen: Hogrefe; 1997. https://doi.org/10.1026//0084-5345.28.1.68.
- [Result] Raven J. Raven´s Progressive Matrices 2, Clinical Edition. 1st ed. München: Pearson; 2019.
- [Result] Gutierrez PM, Osman A, Barrios FX, Kopper BA. Development and initial validation of the Self-harm Behavior Questionnaire. J Pers Assess. 2001 Dec;77(3):475-90. doi: 10.1207/S15327752JPA7703_08. PMID 11781034
- [Result] Wolf M, Limberger MF, Kleindienst N, Stieglitz RD, Domsalla M, Philipsen A, Steil R, Bohus M. [Short version of the borderline symptom list (BSL-23): development and psychometric evaluation]. Psychother Psychosom Med Psychol. 2009 Aug;59(8):321-4. doi: 10.1055/s-0028-1104598. Epub 2009 Mar 9. German. PMID 19274605
- [Result] Lovibond SH, Lovibond PF. Manual for the Depression Anxiety & Stress Scales. 2nd ed. Sydney: Psychology Foundation; 1995.
- [Result] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Result] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Result] EuroQol Research Foundation. EQ-5D-5L User Guide Version 3.0: Basic information on how to use the EQ-5D-5L instrument. Https://EuroqolOrg/Publications/User-Guides 2019.
- [Result] Kuyken W, Hayes R, Barrett B, Byng R, Dalgleish T, Kessler D, Lewis G, Watkins E, Brejcha C, Cardy J, Causley A, Cowderoy S, Evans A, Gradinger F, Kaur S, Lanham P, Morant N, Richards J, Shah P, Sutton H, Vicary R, Weaver A, Wilks J, Williams M, Taylor RS, Byford S. Effectiveness and cost-effectiveness of mindfulness-based cognitive therapy compared with maintenance antidepressant treatment in the prevention of depressive relapse or recurrence (PREVENT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):63-73. doi: 10.1016/S0140-6736(14)62222-4. Epub 2015 Apr 20. PMID 25907157
- [Result] Stiglmayr C, Schmahl C, Bremner JD, Bohus M, Ebner-Priemer U. Development and psychometric characteristics of the DSS-4 as a short instrument to assess dissociative experience during neuropsychological experiments. Psychopathology. 2009;42(6):370-4. doi: 10.1159/000236908. Epub 2009 Sep 15. PMID 19752590
- [Result] Marks IM. Behavioural psychotherapy: Maudsley pocket book of clinical management. Wright/IOP Publishing; 1986.
- [Result] Hutsebaut J, Feenstra DJ, Kamphuis JH. Development and Preliminary Psychometric Evaluation of a Brief Self-Report Questionnaire for the Assessment of the DSM-5 level of Personality Functioning Scale: The LPFS Brief Form (LPFS-BF). Personal Disord. 2016 Apr;7(2):192-7. doi: 10.1037/per0000159. Epub 2015 Nov 23. PMID 26595344
- [Result] Spielberger CD. State-Trait Anger Expression Inventory-2 (STAXI-2). Professional Manual. Tampa, FL: Psychological Assessment Resources; 1999.
- [Result] Stangier U, Schuller J, Brahler E. Development and validation of a new instrument to measure social pain. Sci Rep. 2021 Apr 15;11(1):8283. doi: 10.1038/s41598-021-87351-3. PMID 33859226
- [Result] Honecker H, Bertsch K, Spiess K, Krauch M, Kleindienst N, Herpertz SC, Neukel C. Impact of a Mechanism-Based Anti-Aggression Psychotherapy on Behavioral Mechanisms of Aggression in Patients With Borderline Personality Disorder. Front Psychiatry. 2021 Aug 5;12:689267. doi: 10.3389/fpsyt.2021.689267. eCollection 2021. PMID 34421676
- [Result] Bach B, Kerber A, Aluja A, Bastiaens T, Keeley JW, Claes L, Fossati A, Gutierrez F, Oliveira SES, Pires R, Riegel KD, Rolland JP, Roskam I, Sellbom M, Somma A, Spanemberg L, Strus W, Thimm JC, Wright AGC, Zimmermann J. International Assessment of DSM-5 and ICD-11 Personality Disorder Traits: Toward a Common Nosology in DSM-5.1. Psychopathology. 2020;53(3-4):179-188. doi: 10.1159/000507589. Epub 2020 May 5. PMID 32369820
- [Result] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Result] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Result] Roberts NP, Cloitre M, Bisson J, Brewin CR. International trauma interview (ITI) for ICD- 11 PTSD and complex PTSD (Test Version 3.2). 2019.
- [Result] Hutsebaut J, Kamphuis JH, Feenstra DJ, Weekers LC, De Saeger H. Assessing DSM-5-oriented level of personality functioning: Development and psychometric evaluation of the Semi-Structured Interview for Personality Functioning DSM-5 (STiP-5.1). Personal Disord. 2017 Jan;8(1):94-101. doi: 10.1037/per0000197. Epub 2016 Jun 16. PMID 27845529
- [Result] Jensen J, Burlingame G. An item reduction analysis of the Group Questionnaire. Psychotherapy (Chic). 2018 Jun;55(2):144-150. doi: 10.1037/pst0000145. PMID 29863394
- [Result] Bradley MM, Lang PJ. Measuring emotion: the Self-Assessment Manikin and the Semantic Differential. J Behav Ther Exp Psychiatry. 1994 Mar;25(1):49-59. doi: 10.1016/0005-7916(94)90063-9. PMID 7962581
- [Result] Kasper LA, Hauschild S, Berning A, Holl J, Taubner S. Development and validation of the Mentalizing Emotions Questionnaire: A self-report measure for mentalizing emotions of the self and other. PLoS One. 2024 May 6;19(5):e0300984. doi: 10.1371/journal.pone.0300984. eCollection 2024. PMID 38709789
- [Result] Ehrenthal JC, Zimmermann J, Brenk-Franz K, Dinger U, Schauenburg H, Brahler E, Strauss B. Evaluation of a short version of the Experiences in Close Relationships-Revised questionnaire (ECR-RD8): results from a representative German sample. BMC Psychol. 2021 Sep 14;9(1):140. doi: 10.1186/s40359-021-00637-z. PMID 34521473
- [Result] Kendall PC, Howard BL, Hays RC. Self-Referent Speech and Psychopathology: The Balance of Positive and Negative Thinking 1989;13:583-98. https://doi.org/10.1007/BF01176069.
- [Result] Bateman A, Fonagy P. Mentalization-Based Treatment for Personality Disorders: A practical guide. Oxford: Oxford University Press; 2016.
- [Result] Hilsenroth MJ, Blagys MD, Ackerman SJ, Bonge DR, Blais MA. Measuring Psychodynamic-Interpersonal and Cognitive-Behavioral Techniques: Development of the Comparative Psychotherapy Process Scale. Psychotherapy: Theory, Research, Practice, Training 2005;42:340-56.
- [Result] Talia A, Muzi L. Therapist Attunement Scales Coding System (Unpublished Manuscript). University of Heidelberg 2017.
- [Result] Eubanks CF, Muran JC, Safran J. Rupture Resolution Rating System (3RS): Manual. New York: Unpublished manuscript, Mount Sinai-Beth Israel Medical Center; 2015.
- [Result] Talia A, Miller-Bottome M. Patient Attachment Coding System, 2.0 (Unpublished manuscript). Deparment of Psychology: University of Copenhagen 2012.
- [Result] Rozental A, Kottorp A, Forsstrom D, Mansson K, Boettcher J, Andersson G, Furmark T, Carlbring P. The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother. 2019 Sep;47(5):559-572. doi: 10.1017/S1352465819000018. Epub 2019 Mar 15. PMID 30871650
- [Result] Krause Jacob M, Abarzúa M, Silva M, Navarro D, Altimir Colao C. Psychotherapie aus der Sicht von Klienten mit Schizophrenie. Verhaltenstherapie & Psychosoziale Praxis 2016;47:63-76.
- [Result] Loranger AW, Janca A, Sartorius N. Assessment and diagnosis of personality disorders: The ICD-10 international personality disorder examination (IPDE). Cambridge University Press; 1997.
- [Result] Hatcher RL, Gillaspy JA. Development and validation of a revised short version of the Working Alliance Inventory. Psychotherapy Research. 2006; 16: 12-25.
- [Result] Huber J, Nikendei C, Ehrenthal JC, Schauenburg H, Mander J, Dinger U. Therapeutic Agency Inventory: Development and psychometric validation of a patient self-report. Psychother Res. 2019 Oct;29(7):919-934. doi: 10.1080/10503307.2018.1447707. Epub 2018 Mar 20. PMID 29557306
- [Result] Muller S, Wendt LP, Zimmermann J. Development and Validation of the Certainty About Mental States Questionnaire (CAMSQ): A Self-Report Measure of Mentalizing Oneself and Others. Assessment. 2023 Apr;30(3):651-674. doi: 10.1177/10731911211061280. Epub 2021 Dec 14. PMID 34905983
- [Result] Campbell C, Tanzer M, Saunders R, Booker T, Allison E, Li E, O'Dowda C, Luyten P, Fonagy P. Development and validation of a self-report measure of epistemic trust. PLoS One. 2021 Apr 16;16(4):e0250264. doi: 10.1371/journal.pone.0250264. eCollection 2021. PMID 33861805
- [Result] Gratz KL, Roemer L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. J Psychopathol Behav Assess. 2004; 26: 41-54. https://doi.org/10.1023/B:JOBA.0000007455.08539.94.
- [Derived] Hauschild S, Taubner S, Vidalon Blachowiak T, Dinger U, Gundel H, Herpertz SC, Rademacher J, Strauss B, Storck T, Vassileva R, Burghaus I, Herbst M, Chen S, Nikendei C, Euler S, Volkert J. Mentalization-based treatment versus bona fide treatment for patients with borderline personality disorder in Germany (MAGNET): study protocol of a prospective, multi-centre randomized controlled trial. BMC Psychiatry. 2025 Apr 11;25(1):367. doi: 10.1186/s12888-025-06809-0. PMID 40217262